CLINICAL TRIAL: NCT04614779
Title: Phase IIa Clinical Study to Assess the Safety and Efficacy of CN128 Tablets in the Treatment of Iron Overload in Transfusion Dependent Thalassemia Patients Aged 16 and Above
Brief Title: Long-term Clinical Study of CN128 in Thalassemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Zede Pharma-Tech Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A160605
Record Dates: First submitted 2020-09-23; First posted 2020-11-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Thalassemia; Iron Overload
MeSH Terms: conditions — Thalassemia; Iron Overload

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CN128 Group (Experimental): All subjects will be given the lower (10 mg/kg bw, bid) or higher dose (15 mg/kg bw, bid) for 24 or 48 weeks, according to the administration plan.
  All subjects will be given the lower (15 mg/kg bw, bid) or higher dose (20 mg/kg bw, bid) for 49 or 96 weeks, according to the administration plan.
  The dosage form is tablets.
  Interventions: Drug: CN128 Tablets

INTERVENTIONS:
Drug: CN128 Tablets — Iron chelator, oral tablets
  Other Names: CN128

SUMMARY:
1. Primary objectives:

   • To evaluate the safety and efficacy of long-term orally administration of CN128 in thalassaemia patients with blood transfusion dependent and aged 16 and above.
2. Design:

   * The study is designed as a single arm and opened phase IIa clinical trial, so as to investigate the safety and efficacy of CN128.
   * A total of 50 eligible subjects are planned to be enrolled, and orally administration of CN128 for 24 weeks or 48 weeks according to the administration plan. The treatment period is from day 0 to 24 weeks, and the extended treatment period was from 25 weeks to 96 weeks.
   * Subjects' medication status, uncomfortable symptoms, concomitant medication or non-drug therapy were recorded daily.
3. Subject inclusion criteria:

   * Thalassemia patients.
   * The number of blood transfusion per month ≥1. Or hemoglobin can not be maintained at 90g/L above, if blood transfusions is less than once per month.
   * Serum ferritin ≥ 500 µg/L
   * Patients aged 16 and above
   * Volunteer for the trial and sign the informed consent.
4. Subject exclusion criteria:

   * Active hepatitis B (HBsAg positive, HBsAb negative) or hepatitis C (HCV antibody positive, detectable HCV RNA, and alanine transaminase (ALT) beyond normal range)
   * Active gastrointestinal disease history (including: gastric ulcer, duodenal ulcer, stomach or esophageal varices, ulcerative colitis, Crohn's disease, gastrointestinal cancer, familial genetic multiple intestinal polyps), and History of gastrointestinal perforation, gastrointestinal surgery that influence drug absorption, and other potential intestinal complications considered by researchers;
   * ALT or Aspartate transaminase (AST) > 2.5 × Upper limit of normal (ULN), or serum creatinine > 1.5 × ULN;
   * Neutropenia patient (neutrophil count < 1.5 × 109 / L);
   * Active infection uncontrolled;
   * The patients who are currently taking CYP3A strong inducer or strong inhibitor drugs, or the drug that may extend the QT interval, or the drug that may decrease neutrophil count, but can not temporarily interrupt the use of such drugs;
   * Congenital long QT syndrome or known family history of long QT syndrome; QTc > 480 ms; clinically significant ventricular or atrial fast arrhythmia;
   * The patients who can not accept MRI as detection means, such as claustrophobic for MRI, pacemaker, and those using ferromagnetic metal implants.
   * Birth planner (including male subjects) within or within 3 months after the end of the trial;
   * Participated in other clinical trials in the three months before taking the test preparation, except for non-interventional studies;
   * Pregnant or lactating women;
   * Unsuitable to participate in the trial considered by the researchers.
5. Usage:

   * All subjects will be given the lower (10 mg/kg bw, bid) or higher dose (15 mg/kg bw, bid) for 24 or 48 weeks, according to the administration plan.
   * All subjects will be given the lower (15 mg/kg bw, bid) or higher dose (20 mg/kg bw, bid) for 49 or 96 weeks, according to the administration plan.
6. Safety assessments:

   Safety evaluations include adverse events, adverse reactions, severe adverse events, and severe adverse reactions; growth (weight, height); total and free testosterone in men, follicle-generating hormone and luteinizing hormone in women; vital signs and electrocardiogram; hearing, laboratory tests (blood routine analytes, blood biochemistry, coagulation function, thyroid and para-thyroid function, urine routine analytes.), urine pregnancy test (women of childbearing age),Levels of drug exposure during the study.
7. Efficacy assessments:

   Efficacy evaluations include serum ferritin, liver iron content (MRI R2) and cardiac iron content (MRI T2*).
8. Statistics:

   * Subject characteristic distribution Demographic characteristics, general conditions, and baseline conditions (pre-treatment) of enrolled subjects were analyzed.The measurement data are described by means, standard deviation, minimum value and maximum value, while the qualitative data list frequency and percentage.
   * Safety analysis Descriptive statistical analysis was used for safety endpoints.
   * Effectiveness analysis Mean, standard deviation, median, minimum and maximum values were described and 95% confidence intervals were calculated. Paired T-test was used to compare each time point with the baseline if necessary. The 95% confidence interval was calculated by using Clopper-Pearson method for the proportion of patients.

DETAILED DESCRIPTION:
Clinical Trial - IIa - Study Description - Detailed Description

1. Primary objectives:

   * To evaluate the adverse events, adverse reactions, severe adverse events and severe adverse reactions during the study period, so as to investigate the safety;
   * To evaluate the changes of serum ferritin over time after orally administration of CN128 in thalassaemia patients with blood transfusion dependent and aged 16 and above, so as to investigate the efficacy;
   * To evaluate the effect on iron excretion in liver after orally administration of CN128 for 12, 24 weeks in thalassaemia patients with blood transfusion dependent and aged 16 and above, so as to investigate the efficacy;
   * To evaluate the effect on iron excretion in heart after orally administration of CN128 for 12, 24 weeks in thalassaemia patients with blood transfusion dependent and aged 16 and above, so as to investigate the efficacy;
   * To evaluate the proportion of patients with decreased or unchanged liver iron content after orally administration of CN128 for 12, 24 weeks in thalassaemia patients with blood transfusion dependent and aged 16 and above, so as to investigate the efficacy;
   * To evaluate the safety and efficacy of long-term orally administration of CN128 in thalassaemia patients with blood transfusion dependent and aged 16 and above.
2. Design:

   * The study is designed as a single arm and opened phase IIa clinical trial, so as to investigate the safety and efficacy of CN128.
   * A total of 50 eligible subjects are planned to be enrolled, and orally administration of CN128 for 24 weeks or 48 weeks according to the administration plan. The treatment period is from day 0 to 24 weeks, and the extended treatment period was from 25 weeks to 96 weeks.
   * Administration plan:

   (1)0 day~48 weeks： The trial will start with the lower dose of CN128 (10 mg/kg body weight [bw], bid) for two weeks, then the subjects will return to the study center. If no unacceptable toxicity associated with CN128 is found, the subjects will be given the higher dose (15 mg/kg body weight [bw], bid). If unacceptable toxicity associated with CN128 is found, the subjects will be suspended or stopped administration. If the adverse event turns to normal or abnormal but no clinical significance after suspension administration, the subjects will be given the lower dose of CN128 (10 mg/kg body weight [bw], bid).

   After taking CN128 at 15 mg/kg, if unacceptable toxicity associated with CN128 is found, the dosage will be reduce to 10 mg/kg. If no symptoms appear, the dose can be increased to 15 mg/kg. If the unacceptable toxicity related to CN128 still occurs, the subjects will be suspended or stopped administration. If the adverse event turns to normal or abnormal but no clinical significance after suspension administration, the subjects will be given the lower dose of CN128 (10 mg/kg body weight [bw], bid). The dose will be assessed once every two or four weeks.

   Subjects' medication status, uncomfortable symptoms, concomitant medication or non-drug therapy were recorded daily.

   (2)49 weeks~96 weeks： Subjects who have completed 48 weeks of treatment may continue dosing at the original dose until the end of the study or withdraw early if they do not experience intolerable toxicity associated with CN128 tablets and have fair efficacy (≥20% elevation on MRI T2*) and if, in the judgment of the investigator, the benefits outweigh the risks.

   Subjects who have completed 48 weeks of treatment, who have not experienced intolerable toxicity associated with CN128 tablets, but who have been assessed by the investigator as having poor efficacy (<20% elevation of MRI T2*) and in the judgment of the investigator the benefit outweighs the risk, may, with the subject's consent, have the dosage increased at the additional visit or the established most recent visit to 15 mg/kg in the morning and 20 mg/kg in the evening, with an assessment made at 2 weeks of dosing：

   If no relevant intolerable toxicity occurs, the dose may continue to be increased to 20 mg/kg bid and assessed after 2 weeks of dosing:
   1. If no relevant intolerable toxicity occurs, the 20 mg/kg bid dose may be administered until the end of the study or early withdrawal (daily dose 40 mg/kg/d);
   2. If relevant intolerable toxicity occurs, the dose may be reduced to 15 mg/kg in the morning and 20 mg/kg bid in the evening until the end of the study or early withdrawal (daily dose 35 mg/kg/d).

   If relevant intolerable toxicity occurs, the dose may be reduced to 15 mg/kg bid until the end of the study or early withdrawal (daily dose 30 mg/kg/d).
3. Subject inclusion criteria:

   * Thalassemia patients.
   * The number of blood transfusion per month ≥1. Or hemoglobin can not be maintained at 90g/L above, if blood transfusions is less than once per month.
   * Serum ferritin ≥ 500 µg/L
   * Patients aged 16 and above
   * Volunteer for the trial and sign the informed consent.
4. Subject exclusion criteria:

   * Active hepatitis B (HBsAg positive, HBsAb negative) or hepatitis C (HCV antibody positive, detectable HCV RNA, and ALT beyond normal range)
   * Active gastrointestinal disease history (including: gastric ulcer, duodenal ulcer, stomach or esophageal varices, ulcerative colitis, Crohn's disease, gastrointestinal cancer, familial genetic multiple intestinal polyps), and History of gastrointestinal perforation, gastrointestinal surgery that influence drug absorption, and other potential intestinal complications considered by researchers;
   * ALT or AST > 2.5 × ULN, or serum creatinine > 1.5 × ULN;
   * Neutropenia patient (neutrophil count < 1.5 × 109 / L);
   * Active infection uncontrolled;
   * The patients who are currently taking CYP3A strong inducer or strong inhibitor drugs, or the drug that may extend the QT interval, or the drug that may decrease neutrophil count, but can not temporarily interrupt the use of such drugs;
   * The patients who are allergic or contraindicated to the main ingredients or excipients of CN128 tablets;
   * Congenital long QT syndrome or known family history of long QT syndrome; QTc > 480 ms; clinically significant ventricular or atrial fast arrhythmia;
   * The patients who can not accept MRI as detection means, such as claustrophobic for MRI, pacemaker, and those using ferromagnetic metal implants;
   * Birth planner (including male subjects) within or within 3 months after the end of the trial;
   * Participated in other clinical trials in the three months before taking the test preparation, except for non-interventional studies;
   * Pregnant or lactating women;
   * Unsuitable to participate in the trial considered by the researchers.
5. Usage:

   All subjects will be given the lower (10 mg/kg bw, bid) or higher dose (15 mg/kg bw, bid) for 24 or 48 weeks, according to the administration plan.

   All subjects will be given the lower (15 mg/kg bw, bid) or higher dose (20 mg/kg bw, bid) for 49 or 96 weeks, according to the administration plan.
6. Safety assessments:

   Safety evaluations include adverse events, adverse reactions, severe adverse events, and severe adverse reactions; growth (weight, height); total and free testosterone in men, follicle-generating hormone and luteinizing hormone in women; vital signs and electrocardiogram; hearing, laboratory tests (blood routine analytes, blood biochemistry, coagulation function, thyroid and para-thyroid function, urine routine analytes.), urine pregnancy test (women of childbearing age),Levels of drug exposure during the study.
7. Efficacy assessments:

   Efficacy evaluations include serum ferritin, liver iron content (MRI R2) and cardiac iron content (MRI T2*).
8. Statistics:

   * Subject characteristic distribution Demographic characteristics, general conditions, and baseline conditions (pre-treatment) of enrolled subjects were analyzed.The measurement data are described by means, standard deviation, minimum value and maximum value, while the qualitative data list frequency and percentage.
   * Safety analysis Descriptive statistical analysis was used for safety endpoints. Summarize the incidence of adverse events, adverse reactions, adverse events leading to withdrawal from the trial, adverse events leading to death, severe adverse events, and severe adverse reactions. The incidence is calculated by subsystem, symptom/sign. Severity of adverse events and adverse reactions: if multiple adverse events occur in the same subject, the most serious one is included in the analysis; if different adverse events occurred in the same subject, the most severe adverse events were counted in the analysis. Drug exposure during the study: describe medication compliance during the study, actual dose, administration adjustments during the study, whether the study was discontinued, and reasons for the suspension.
   * Effectiveness analysis Mean, standard deviation, median, minimum and maximum values were described and 95% confidence intervals were calculated. Paired T-test was used to compare each time point with the baseline if necessary. The 95% confidence interval was calculated by using Clopper-Pearson method for the proportion of patients.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia patients.
* The number of blood transfusion per month ≥1. Or hemoglobin can not be maintained at 90g/L above, if blood transfusions is less than once per month.
* Serum ferritin ≥ 500 µg/L
* Patients aged 16 and above
* Volunteer for the trial and sign the informed consent.

Exclusion Criteria:

* Active hepatitis B (HBsAg positive, HBsAb negative) or hepatitis C (HCV antibody positive, detectable HCV RNA, and ALT beyond normal range)
* Active gastrointestinal disease history (including: gastric ulcer, duodenal ulcer, stomach or esophageal varices, ulcerative colitis, Crohn's disease, gastrointestinal cancer, familial genetic multiple intestinal polyps), and History of gastrointestinal perforation, gastrointestinal surgery that influence drug absorption, and other potential intestinal complications considered by researchers;
* ALT or AST > 2.5 × ULN, or serum creatinine > 1.5 × ULN;
* Neutropenia patient (neutrophil count < 1.5 × 109 / L);
* Active infection uncontrolled;
* The patients who are currently taking CYP3A strong inducer or strong inhibitor drugs, or the drug that may extend the QT interval, or the drug that may decrease neutrophil count, but can not temporarily interrupt the use of such drugs;
* The patients who are allergic or contraindicated to the main ingredients or excipients of CN128 tablets;
* Congenital long QT syndrome or known family history of long QT syndrome; QTc > 480 ms; clinically significant ventricular or atrial fast arrhythmia;
* The patients who can not accept MRI as detection means, such as claustrophobic for MRI, pacemaker, and those using ferromagnetic metal implants;
* Birth planner (including male subjects) within or within 3 months after the end of the trial;
* Participated in other clinical trials in the three months before taking the test preparation, except for non-interventional studies;
* Pregnant or lactating women;
* Unsuitable to participate in the trial considered by the researchers.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, adverse reactions, severe adverse events and severe adverse reactions as a measure of safety and tolerability during the study period | up to 96 weeks
  To determine the incidence, type and severity of adverse events, adverse reactions, severe adverse events and severe adverse reactions in patients up to 96 weeks.
Absolute Change in Weight (Unit: kg) From Baseline Over Time | Baseline, 24, 48, 72 and 96 weeks.
  The patient's weight will be determined, and it's one kind of Physical examination.
Absolute Change in Height (Unit: m) From Baseline Over Time | Baseline,24, 48, 72 and 96 weeks.
  The patient's height will be determined, and it's one kind of Physical examination.
Absolute Change in Hormon (total and free testosterone in men, follicle-generating hormone and luteinizing hormon in women) From Baseline Over Time | Baseline, 24, 48, 72 and 96 weeks.
  Hormon will be determined, and it's one kind of laboratory test.
Absolute Change in Temperature (Unit: ℃）From Baseline Over Time | Baseline, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's temperature will be determined, and it's one kind of vital signs checks.
Absolute Change in Blood pressure (Unit: mmHg ) From Baseline Over Time | Baseline, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  Both patient's systolic and diastolic blood pressure will be measured, and it's one kind of vital signs checks.
Absolute Change in Heart rate (Unit: bpm) From Baseline Over Time | Baseline, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's heart rate will be determined, and it's one kind of vital signs checks.
Absolute Change in Respiration (Unit: bpm) From Baseline Over Time | Baseline, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's respiration will be determined, and it's one kind of vital signs checks.
Absolute Change in Electrocardiogram (P-R (Unit: ms), QRS (Unit: ms), QTc (Unit: ms), etc) From Baseline Over Time | Baseline, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's electrocardiogram will be measured, and it's one kind of laboratory test.
Change in Auditory Function From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's auditory function will be determined by otorhinolaryngology.
Absolute Change in White Blood Count (Unit: 10E9/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's white blood count will be determined, and it's one kind of laboratory test.
Absolute Change in Neutrophil Count (Unit: 10E9/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's neutrophil count will be determined, and it's one kind of laboratory test.
Absolute Change in Lymphocyte Count (Unit: 10E9/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's lymphocyte count will be determined, and it's one kind of laboratory test.
Absolute Change in Monocyte Count (Unit: 10E9/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's monocyte count will be determined, and it's one kind of laboratory test.
Absolute Change in Eosinophilic Count (Unit: 10E9/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's eosinophilic count will be determined, and it's one kind of laboratory test.
Absolute Change in Basophilic Count (Unit: 10E9/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's basophilic count will be determined, and it's one kind of laboratory test.
Absolute Change in Red Blood Count (Unit: 10E9/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's red blood count will be determined, and it's one kind of laboratory test.
Absolute Change in Hemoglobin (Unit: g/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's hemoglobin will be determined, and it's one kind of laboratory test.
Absolute Change in Hematocrit (Unit:%) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's hematocrit will be determined, and it's one kind of laboratory test.
Absolute Change in Blood Platelet Count (Unit: 10E9/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's blood platelet count will be determined, and it's one kind of laboratory test.
Absolute Change in Thrombocytocrit (Unit: %) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's thrombocytocrit will be determined, and it's one kind of laboratory test.
Absolute Change in Alanine Aminotransferase (Unit: U/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's alanine aminotransferase will be determined, and it's one kind of laboratory test.
Absolute Change in Total Bilirubin (Unit:µmol/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's total bilirubin will be determined, and it's one kind of laboratory test.
Absolute Change in Total Protein (Unit:g/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's total protein will be determined, and it's one kind of laboratory test.
Absolute Change in Albumin (Unit: g/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's albumin will be determined, and it's one kind of laboratory test.
Absolute Change in Globulin (Unit: g/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's globulin will be determined, and it's one kind of laboratory test.
Absolute Change in Alkaline Phosphatase (Unit: U/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's alkaline phosphatase will be determined, and it's one kind of laboratory test.
Absolute Change in Lactate Dehydrogenase (Unit: IU/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's lactate dehydrogenase will be determined, and it's one kind of laboratory test.
Absolute Change in Urea (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's urea will be determined, and it's one kind of laboratory test.
Absolute Change in Creatinine (Unit:µmol/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's creatinine will be determined, and it's one kind of laboratory test.
Absolute Change in Glucose (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's glucose will be determined, and it's one kind of laboratory test.
Absolute Change in Potassium (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's potassium will be determined, and it's one kind of laboratory test.
Absolute Change in Sodium (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's sodium will be determined, and it's one kind of laboratory test.
Absolute Change in Chlorine (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's chlorine will be determined, and it's one kind of laboratory test.
Absolute Change in Calcium (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's calcium will be determined, and it's one kind of laboratory test.
Absolute Change in Aspartate Aminotransferase (Unit: U/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's aspartate aminotransferase will be determined, and it's one kind of laboratory test.
Absolute Change in Fibrinogen (Unit: g/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's fibrinogen will be determined, and it's one kind of laboratory test.
Absolute Change in Prothrombin time (Unit: s) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's prothrombin time will be determined, and it's one kind of laboratory test.
Absolute Change in Activated Partial Thromboplastin Time (APTT, Unit: s) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's APTT will be determined, and it's one kind of laboratory test.
Absolute Change in Thyroid and para-gland function (Serum total thyroxine, parathyroid hormone, total triiodothyronine and thyrotropin) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's thyroid and para-gland function will be determined, and it's one kind of laboratory test.
Absolute Change in Urine Glucose (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's urine glucose will be determined, and it's one kind of laboratory test.
Absolute Change in Urine Protein (Unit: g/L)) From Baseline Over Time | Baseline, 2, 12, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  The patient's urine protein will be determined, and it's one kind of laboratory test.
Absolute Change in Dosage（mg/kg）during the study period | Up to 96 weeks
  The dosages will be investigated up to 96 weeks.
Duration of Administration during the study period | Up to 96 weeks
  The duration of administration will be investigated up to 96 weeks.
Number of Participants during the study period | Up to 96 weeks
  The number of participants will be investigated up to 96 weeks.
Absolute Change in Serum ferritin (Unit: µg/L) From Baseline Over Time | Baseline, 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84 and 96 weeks.
  Serum ferritin will be determined, and it's one kind of laboratory test.
Absolute Change in Liver iron content (MRI R2) From Baseline Over Time | Baseline, 12, 24, 48, 72 and 96 weeks.
  Liver iron content will be determined by liver magnetic resonance.
Absolute Change in Heart iron content (MRI T2*) From Baseline Over Time | Baseline, 12, 24, 48, 72 and 96 weeks.
  Heart iron content will be determined by cardio magnetic resonance.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Jianmin, PhD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital Of Guangxi Medical University, Nanning, Guangxi, China